CLINICAL TRIAL: NCT02346760
Title: A Phase I, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Subcutaneous Dose of UB-621 in Healthy Volunteers
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of UB-621 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United BioPharma (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A101-HSV
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Herpes Simplex Virus Infection
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UB-621 (Experimental): Intervention drug: UB-621
  Interventions: Drug: UB-621

INTERVENTIONS:
Drug: UB-621 — 100 mg/ml, subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of a single subcutaneous dose of UB-621 in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase I, open-label, single dose, dose escalation study in healthy volunteers. Eligible volunteers will be sequentially enrolled into four escalating-dose cohorts at a study site. After administration of a single subcutaneous dose of UB-621, subjects will be followed for 70 or 112 days and monitored for safety, tolerability, and pharmacokinetics parameters.

ELIGIBILITY:
Inclusion Criteria:

* With age between 20 and 55 years.
* With no clinically relevant abnormalities in vital signs, and clinical laboratory tests at screening visit judged by investigator.
* Body weight: <85 kg.
* Subject has signed the written informed consent form.

Exclusion Criteria:

* With significant active infection (acute or chronic) within 28 days prior to the screening visit.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic diseases, or clinical findings within 3 months prior to the screening visit.
* Positive serology for HIV antibody, HCV antibody or HBV surface antigen.
* Female subjects who are breastfeeding, pregnant, and planning to become pregnant during the study period.
* The clinical investigator considers that the subject is not in the condition to participate in this study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 70 or 112 days

SECONDARY OUTCOMES:
Peak concentration of UB-621 | Up to 70 or 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wai Wong, MD, Principal Investigator — Taipei Veterans General Hoapital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan